CLINICAL TRIAL: NCT05781503
Title: Transitioning Youth Out of Homelessness 2.0: a Pilot Randomized Controlled Trial of a Rent Subsidy and Identity Capital Intervention for Youth Exiting Homelessness
Brief Title: Transitioning Youth Out of Homelessness 2.0 (TYOH 2.0)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Covenant House Toronto (Other); StepStones for Youth (Unknown); Living Rock Ministries (Other); Resource Association for Teens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-230
Record Dates: First submitted 2023-02-27; First posted 2023-03-23 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2023-07

CONDITIONS: Homelessness; Youth
Keywords: Identity Capital; Youth; Rent Subsidy; Coach; Self-Efficacy; Self-Esteem; Control; Purpose; Socioeconomic Inclusion; Homelessness; Transition

STUDY DESIGN:
Intervention Model Description: This pilot study will employ a convergent mixed methods (quantitative and qualitative data collected concurrently and the findings combined), two-arm parallel RCT (participants randomly assigned to either one intervention or control group), open-label (participants and research team aware of random assignment) design with 1:1 allocation (roughly equal number of participants in each study arm) embedded within a Community Based Participatory Action Research framework. Twenty young people will be allocated to the intervention group (portable rent subsidies + identity capital intervention), while 20 will be allocated to the control group (portable rent subsidies only). Participants in the intervention group (n = 20) will receive 12 months of: portable rent subsidies, engage in a co-designed (with youth who have experienced homelessness) leadership guide, and be assigned a coach (one coach/10 youth).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Portable Rent Subsidies + Identity Capital Intervention (Experimental): Young people randomized to the intervention group will receive 12 months of: portable rent subsidies, engage in a co-designed leadership guide, and be assigned a coach (one coach/10 youth).
  Interventions: Behavioral: Identity Capital Intervention (Coach + Co-designed Leadership Guide); Other: Monthly Rent Subsidies
- Portable Rent Subsidies Only (Active Comparator): The control group will be offered 12 months of portable rent subsidies.
  Interventions: Other: Monthly Rent Subsidies

INTERVENTIONS:
Behavioral: Identity Capital Intervention (Coach + Co-designed Leadership Guide) — Young people randomized to the intervention group will engage in a co-designed leadership guide with their assigned coach. The co-designed leadership guide contains 12 chapters with the overarching aim of enhancing identity capital along with providing strategies to achieve participant-identified goals. Each chapter contains four activities (e.g., self-reflection exercise or listening to a podcast). Ideally, youth will complete one chapter every month. Each young person in this group will meet individually with their coach every two weeks and with a larger group of 10 youth participants and their coach every month.
  Arms: Portable Rent Subsidies + Identity Capital Intervention
Other: Monthly Rent Subsidies — All study participants will receive a monthly rent subsidy ($800 for those living in Toronto; $700 for those living in St. Catharine's or Hamilton due to differences in cost of living) for 12 months.

SUMMARY:
Introduction: This 12-month pilot randomized controlled trial (RCT) built on previous community-engaged work and explored whether portable rent subsidies and an intervention targeting identity capital (purpose, control, self-efficacy, and self-esteem) hold promise as a way to facilitate socioeconomic inclusion for youth (age 16 - 24 years) exiting homelessness and living in market rent housing in Ontario, Canada. All (n = 40) participants received rent subsidies; half were randomly assigned an identity capital intervention (co-designed leadership guide + coach).

Methods and analysis: This study employed a convergent mixed methods, two-arm parallel RCT, open-label design with 1:1 allocation embedded within a Community Based Participatory Action Research framework and underpinned by Critical Social Theory.

Specifically, the objectives and measures were:

1. Primary - to examine whether targeted economic and identity-based supports are a feasible and acceptable way to foster socioeconomic inclusion. Measures: recruitment/enrolment/dropout metrics; self-report composite checklists regarding intervention engagement; coaching session attendance; qualitative focus groups.
2. Secondary - to assess differences between targeted economic and identity-based supports (intervention group) and economic supports only (control group) at the 12-month primary endpoint with respect to self-reported socioeconomic inclusion measures of: 1) education, employment and training (EET); 2) housing security; and 3) identity capital. Measures: self-report composite EET checklist; self-report measures of housing security and identity capital.
3. Exploratory - to explore whether the estimated effect of the intervention differed by baseline variables or level of engagement with the intervention. Measures: select variables from the baseline demographic questionnaire; GAIN-Short Screener questionnaire for those in the intervention group.

Ethics and dissemination: This study received ethical approval from the Unity Health Toronto Research Ethics Board. The investigators will continue working alongside community partners - including youth with lived expertise - to disseminate findings broadly and in diverse formats.

DETAILED DESCRIPTION:
The overarching aim of this mixed methods study was to determine the feasibility and acceptability of a strengths-based intervention focused on building identity capital, as a way to facilitate socioeconomic inclusion for youth (age 16 - 24 years) exiting homelessness and living in market rent housing.

Specifically, the objectives were to:

1. Primary - examine the feasibility and acceptability of a RCT of targeted economic and identity-based supports to foster socioeconomic inclusion.
2. Secondary - estimate the effect of adding identity-based supports to economic supports (intervention group) compared with economic supports alone (control group) at the 12-month endpoint with respect to self-reported proxy indicators of socioeconomic inclusion.
3. Exploratory - among the intervention group, explore whether the estimated effect of the intervention differs by baseline variables or level of engagement with the intervention.

This pilot study employed a convergent mixed methods (quantitative and qualitative data collected concurrently and the findings combined), two-arm parallel RCT (participants randomly assigned to either the intervention or control group), open-label (participants and research team aware of random assignment) design with 1:1 allocation (equal number of participants in each study arm) embedded within a CBPAR framework.

The study was conducted collaboratively with four community partners who serve youth who are experiencing or have experienced homelessness: 1) Covenant House Toronto (Toronto, ON); 2) Living Rock (Hamilton, ON); 3) The RAFT (St. Catharines, ON); and 4) StepStones for Youth (Toronto, ON). Study participants were recruited from the cities in which our community partners are located: Toronto, ON (Greater Toronto Area population 6.7 million); Hamilton, ON (population 785,000); and St. Catharines, ON (St. Catharines-Niagara population 416,000).

Youth in both arms (n = 40) were provided monthly rent subsidies ($700.00 CAD/month Hamilton and St. Catharines; $800.00 CAD/month Toronto) for 12 months, which was paid directly to landlords and facilitated by our community partners. Youth randomized to the intervention group (n = 20) were also provided a co-designed leadership guide and assigned a study coach. The control group (n = 20) was offered the co-designed leadership guide at the end of the study.

The strengths-based leadership guide - Finding Home: A Guide for Youth in Transition - was co-designed with 12 youth who had experienced homelessness, including youth who participated in TYOH 1.0. The Leadership Guide contained 12 chapters with the overarching aim of enhancing identity capital along with providing strategies to achieve participant-identified goals. Each chapter contained four activities (e.g., self-reflection exercise or listening to a podcast). While the guide was designed for individual study, it was also meant to serve as a reference point for individual and group discussions with the study coaches.

The role of the coach was to speak with youth about how to draw on internal resources to help orient them toward their preferred future. This role was different from case management or mentorship in that a specific coaching methodology (Brief Solution-Focused Coaching) was utilized to walk alongside youth as they developed strategies to reach self-defined goals. Each coach was instructed to devote 2.5 days/week to the intervention and was given a caseload of 9-11 youth. The coaches were instructed to meet individually with each youth on their caseload every two weeks and collectively with the rest of the youth in their group every month.

Questionnaires were completed at baseline. four-, eight-, and 12-months post-randomization. Quantitative analysis was performed using the intention-to-treat principle; that is, all participants were included and analyzed in the groups they were originally randomized. Baseline characteristics of the intervention and control groups were summarized using descriptive statistics (i.e., mean, standard deviation, median and interquartile range for continuous variables, and frequencies and proportions for categorical variables).

Primary outcomes were analyzed by estimating the recruitment rate as the proportion of contacted individuals who expressed interest in participating in the study. The enrollment rate was calculated as the proportion of recruited individuals who were eligible and consented to participate in the study. Dropout rates were separately calculated for intervention and control groups at the end of the study as the 1 - proportion of randomized participants who completed the study at 12 months. Exact (Clopper-Pearson) 95% confidence limits were also calculated.

Secondary outcomes were analyzed by calculating descriptive statistics at each study time point and exploring differences in trajectories from baseline to 12 months follow-up between intervention and control groups using scatterplots and box-plots. Adjusted mean group differences with 95% confidence intervals in continuous outcomes at 12 months (housing security and identity capital) between participants who received the intervention and control participants were estimated using analysis of covariance (i.e., linear regression models), including an indicator of intervention group and the baseline value of the outcome, adjusting for site. We performed regression diagnostics and repeated analyses using the non-parametric Wilcoxon rank-sum test if there were extreme outliers or influential observations.

Exploratory sub-group analysis was conducted considering only the intervention group and stratifying the primary outcomes by selected baseline demographics (for example, gender) or severity levels of components of the Global Appraisal of Individual Needs Short Screener (GAIN-SS) V.3.0.2. We also calculated the correlation between secondary outcomes and the level of engagement with the intervention measured as the percentage of class sessions attended out of a maximum of 24 over the 12-month period. Spearman correlation and Spearman partial correlation coefficients were calculated.

Focus groups with those in the intervention group was conducted at four-, eight-, and 12-months post-randomization. Focus group questions primarily centred around intervention acceptability but also explored the impact of the intervention on identity capital and socioeconomic inclusion (e.g., connection to broader social networks). Analysis began during and after the first data generation session, meaning the questions asked evolved over time based on our preliminary interpretations of the data.

Working alongside community partners to disseminate findings with the aim of highlighting sociostructural inequities, building community capacity, and improving the lives of the youth we serve is fundamental to this work. We anticipate disseminating our findings broadly to community-based and academic audiences in a variety of formats ranging from oral presentations to scientific journal papers.

ELIGIBILITY:
Eligible young people ages 16 - 24 years who have left homelessness within the past 12 months and are currently living or planning to live in market rent housing will be identified by the community partners. This age mandate was chosen because this is the age group served by the community partners. The investigators have chosen to target the first year of exiting homelessness because their collective experience has shown that this is a particularly precarious time for youth in terms of mental health challenges and risk of returning to homelessness.

Inclusion Criteria:

* Be able to provide free and informed consent.
* Be able to understand English (intervention and data collection will be conducted in English).
* Have experienced homelessness (e.g., all non-parental and unstable housing arrangements including shelter stays, couch surfing, and time-limited housing) in the past 12 months.
* Be willing to actively participate in the intervention (co-designed leadership program + coach) if randomized to this arm.

Exclusion Criteria:

* In imminent danger of losing their housing and not able to utilize the rent subsidy to sustain market rent housing.
* Currently receiving rent subsidies.
* Enrolled in a program or study with similar features to the TYOH 2.0 intervention.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Change in intervention feasibility and acceptability as assessed by recruitment/enrolment/dropout metrics from baseline to 12-months. | Assessed at baseline and 12-months.
  To examine intervention feasibility and acceptability, quantitative measures consisting of recruitment/enrolment/dropout metrics will be utilized. Recruitment rate will be estimated as the proportion of contacted individuals who express interest in participating in the study. The enrollment rate will be calculated as the proportion of recruited individuals who are eligible and consent to participate in the study. Dropout rates will be separately calculated for intervention and control groups at the end of the study as the 1 - proportion of randomized participants who completed the study at 12 months. Exact (Clopper-Pearson) 95% confidence limits will also be calculated.
Change in intervention feasibility and acceptability as assessed by the Intervention Engagement Questionnaire from 4-months to 12-months, and coaching session attendance measured across the entire 12-month period. | Assessed at 4-months, 8-months, and 12-months.
  Initially, the study was designed to assess changes in intervention feasibility and acceptability using the Intervention Engagement Questionnaire. This five-item self-report measure was developed for this study and explores engagement with the co-designed leadership guide and coaching (administered only to intervention participants). Higher scores indicate greater engagement.
  However, as the study progressed, we shifted focus to coaching session attendance, as recorded by coaches. Among those in the intervention group, acceptability was measured as the percentage of coaching sessions attended over the 12-month period, out of a maximum of 24 sessions. This provides an objective measure of participant engagement, as self-reported engagement data is not included in the analysis.
Intervention feasibility and acceptability as informed by focus groups from 4-months to 12-months. | Assessed at 4-months, 8-months, and 12-months.
  Focus group questions explored intervention feasibility and acceptability.

SECONDARY OUTCOMES:
Mean change from baseline in housing security as measured by the Housing Security Scale at 12-months. | Assessed at baseline, 4-months, 8-months, and 12-months.
  This 20-item self-report measure explores domains related to: housing need; subjective stability; safety net; threats to stability. Score range: 20-120; higher scores indicate more housing security (internal consistency for subjective stability sub-scale α = 0.71; other sub-scales have not been validated).
Mean change from baseline in identity capital as measured by the Multi-Measure Agentic Personal Scale (MAPS20) at 12-months. | Assessed at baseline, 4-months, 8-months, and 12-months.
  This 20-item validated self-report measure explores domains related to identity capital: self-esteem; purpose in life; internal locus of control; self-efficacy/ego strength. Score range: 20-120; score of less than 71 indicates risk/vulnerability of being overwhelmed by any adverse circumstances (internal consistency of four sub-scales α = .61-.75).
Change in employment, education, and training as assessed by a questionnaire from baseline to 12-months. | Assessed at baseline and 12-months.
  This five-item self-report measure was developed for this study and explores engagement in education (secondary or post-secondary), employment (full- or part-time; formal and informal), and training (paid or unpaid apprenticeship). Employment, education, and training (EET) is a composite binary outcome, where EET = 1 if participants are attending classes, employed, or participating in a training program, and EET = 0 otherwise.

OTHER OUTCOMES:
Subgroup feasibility and acceptability as measured by the Baseline Demographic Questionnaire. | Assessed at baseline.
  This 17-item self-report measure was developed for this study and explores domains related to: age; gender; race/ethnicity; sexual orientation; immigration status; child welfare involvement; homelessness entrenchment; education; social support; financial support; physical health support; mental health support; food security.
Subgroup feasibility and acceptability as measured by the GAIN Short Screener (GAIN-SS). | Assessed at baseline.
  This 23-item validated self-report measure explores: internalizing disorders (e.g., anxiety/depression); externalizing disorders (e.g., impulsivity/disruptive conduct; substance disorders (e.g., illicit drug/alcohol abuse); and crime and violence (e.g., illegal activities/fighting). Severity levels are: 0 problems = low (unlikely to have a diagnosis or need services); 1-2 problems = moderate (a possible diagnosis; the client is likely to benefit from a brief assessment); 3 or more problems = high (high probabilities of a diagnosis; the client is likely to need more formal assessment and intervention, either directly or through referral).
Correlation between secondary outcomes and engagement with the intervention. | Assessed at 12-months.
  The correlation between secondary outcomes and the level of engagement with the intervention (measured as the percentage of coaching sessions attended out of a maximum of 24 over the 12-month period) was explored using Spearman correlation and Spearman partial correlation coefficients.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi S Thulien, NP-PHC, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thulien NS, Stark RK, Amiri A, Abramovich A, Akdikmen A, Carasco A, Daley M, Downey B, Fambegbe OP, Frederick T, Hwang SW, Kozloff N, Noble A, Pedersen C, Rampersaud M, Rodney R, Tibebu T, Nisenbaum R. A Rent Subsidy and Identity Capital Intervention for Youth Exiting Homelessness: Protocol for the Transitioning Youth Out of Homelessness 2.0 Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 25;14:e66210. doi: 10.2196/66210. PMID 40279147
- See also: TYOH 1.0 study website (includes short documentary and animation of study findings). — http://www.searchingforhome.ca